CLINICAL TRIAL: NCT00599794
Title: A Simple Clinical Tool to Help Assess Patient Volume (Fluid) Status
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Allina Health System (Other)
Responsible Party: A. Scott Keller, Mayo Clinic
Other Study IDs: 05-004138
Record Dates: First submitted 2008-01-11; First posted 2008-01-24 (Estimated); Last update posted 2008-01-24 (Estimated); Status verified 2008-01

CONDITIONS: Sepsis
Keywords: Sepsis; Intravascular volume; Ultrasound; Noninvasive measurement
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Healty volunteers who are euvolemic.
- 2: Critically ill patients who will be having a central venous catheter with a monitor to measure central venous pressure placed as part of their planned care independent of this study.

SUMMARY:
Patients may have actual or relative intravascular volume depletion in a number of different disease states, particularly with sepsis syndrome. However, it is clinically difficult to determine volume status without invasive monitoring, which may cause unintended complications. Our hypothesis is that we can accurately estimate central venous pressure, which is a surrogate marker of volume status, with a noninvasive portable ultrasound device.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older.
* Healthy, euvolemic volunteers and critically ill patients who are already in an intensive care unit and who will have a central venous catheter placed as part of their planned medical treatment.

Exclusion Criteria:

* Inability to use ultrasound to measure jugular vein (neck brace or bandage), "code" situation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers, then critically ill patients already in the intensive care unit who are felt to have intravascular volume depletion.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2006-01; Primary Completion 2007-10 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: A. S. Keller, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota